CLINICAL TRIAL: NCT02234765
Title: Management of Patients With Suspected Sleep Apnea Syndrome From Primary Care: Territorial Assistance Network.
Brief Title: Management of Patients With Suspected of Sleep Apnea-hypopnea Syndrome From Primary Care
Acronym: GESAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Ferran Barbe, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PI13/02004
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Sleep Apnea Syndrome
Keywords: OSA; OSAS; Sleep apnea; Management; Primary Care; Sleep Unit; Cost-Effectiveness; ESS
MeSH Terms: conditions — Sleep Apnea Syndromes

ARMS (2):
- Sleep Unit (Active Comparator): Patients diagnosed and followed up in the Sleep Unit.
  Interventions: Other: Standard management
- Primary Care (Experimental): Patients diagnosed and followed up in the Primary Care.
  Interventions: Other: Primary Care-based management

INTERVENTIONS:
Other: Primary Care-based management — Patients will be diagnosed and follow-up in Primary Care.
  Arms: Primary Care
Other: Standard management — Standard management according to Spanish Respiratory Society guidelines in Sleep Unit.
  Arms: Sleep Unit

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is characterized by the manifestation of excessive sleepiness secondary to repeated obstruction of the upper airway during sleep and cognitive-behavioral, respiratory, cardiac, metabolic or inflammatory disorders. Epidemiological studies in our country have shown that OSA is a highly prevalent disease in the general population, affecting 2-4% of the adult population. The most important clinical manifestations of OSAS is a deterioration in the quality of life and an increase in cardiovascular disease. OSA is also associated with traffic accidents. Therefore, and considering the medical complications of OSA, as well as the sociolaboral impact and its negative impact on quality of life and survival; is stated that this disease is a public health problem that requires the physician to identify patients eligible to treatment. Moreover, it has been shown that undiagnosed patients, duplicate the consumption of health resources, comparing when the diagnosis and treatment has been established. Finally, we have a highly effective treatment using positive pressure in the upper airway (CPAP) that has been shown to be effective and cost-effective. The current situation in which all patients diagnosed with OSA and receiving different treatments are monitored and controlled by the Sleep Units (SU) is an oversized medicine specialist at the expense of primary care (PC). Our working hypothesis is: "By the coordination of actions at various levels including interactive training equipment AP, use the bilateral (SU-AP) of electronic medical records and the use of new technologies can be achieved in AP satisfactory management of the diagnostic and therapeutic process of patients with suspected OSA. Patients assisted in both areas have a level of clinical response, satisfaction, compliance and avoidance of complications, similar to that obtained with monitoring by SU. In addition, management by AP will be more cost-effective than in the SU."

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old
* Suspected OSA patients (chronic snoring, apneas, excessive daytime sleepiness) or resistant hypertension
* Written informed consent signed

Exclusion Criteria:

* Patients with impaired lung function (sd. overlap, obesity hypoventilation, and restrictive disorders)
* Severe heart failure
* Severe chronic pathology associated
* Psychiatric disorder
* Periodic leg movements
* Pregnancy
* Other dyssomnias or parasomnias
* Patients already treated with CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in daytime sleepiness (ESS score) at 6 months | baseline and 6 months
  Epworth Sleepiness Scale (ESS)
Cost-effectiveness at 6 months | 6 months
  QUALYS

SECONDARY OUTCOMES:
Change from baseline in quality of life | baseline and 6 months
  EuroQol (EQ5D)
Satisfaction at 6 months | 6 months
  Visual analog scale
CPAP compliance at 6 months | 6 months
  Objective data to be downloaded from the CPAP device
Adverse events at 6 months | 6 months
  Adverse events / secondary effects related to CPAP compliance.
Change from baseline in blood pressure | Baseline and 6 months
  Office blood pressure
Change from baseline in body mass index | Baseline and 6 months
Lost of follow up / Abandons at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbe, MD, Principal Investigator — Hospital Arnau de Vilanova. IRB Lleida. CIBERes
Locations (1):
- Hospital Arnau de Vilanova-Santa María, Lleida, Lleida, Spain

REFERENCES:
- [Derived] Tarraubella N, Sanchez-de-la-Torre M, Nadal N, De Batlle J, Benitez I, Cortijo A, Urgeles MC, Sanchez V, Lorente I, Lavega MM, Fuentes A, Clotet J, Llort L, Vilo L, Juni MC, Juarez A, Gracia M, Castro-Grattoni AL, Pascual L, Minguez O, Masa JF, Barbe F. Management of obstructive sleep apnoea in a primary care vs sleep unit setting: a randomised controlled trial. Thorax. 2018 Dec;73(12):1152-1160. doi: 10.1136/thoraxjnl-2017-211237. Epub 2018 Jul 31. PMID 30064993